CLINICAL TRIAL: NCT05269875
Title: Advance Care Planning in Patients With Heart Failure in Denmark (DanHFacp): a Study Protocol
Brief Title: Advance Care Planning in Patients With Heart Failure in Denmark
Acronym: DanHFacp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Southern Denmark (Other); Odense University Hospital (Other); Zealand University Hospital (Other); REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other)
Responsible Party: Principal Investigator, Camilla Charlotte Lykke, Principal Investigator, Postdoc, Nordsjaellands Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ACP-P-2020-790
Record Dates: First submitted 2022-02-02; First posted 2022-03-08 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Heart Failure; Advance Care Planning; Communication; Feasibility Studies
Keywords: Heart Failure; Advance care planning; Feasibility study; Adaptation; Complex intervention; Communication
MeSH Terms: conditions — Heart Failure; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advance care planning in heart failure patients (Other): The patient and their closest relative will be offered a palliative care intervention by the Department of Cardiology.
  Interventions: Other: ACP

INTERVENTIONS:
Other: ACP — The intervention covers a formal ACP discussion, including provision of a holistic approach (physical, psychological, spiritual, social) and includes symptom control and discussion on illness limitations and prognosis, goal assessment and goal adjustment, financial issue, (un)desirable treatments for current and future care, hopes and wishes, and possibility of involvement of a palliative care team.

SUMMARY:
Advance care planning (ACP) represents a process whereby a patient, in consultation with healthcare professionals, family members and important others, makes decisions about his or her future healthcare and wishes for end-of-life care and is widely advocated to improve end-of-life care for patients with heart failure (HF). Despite the growing emphasis on communication with HF patients and their relatives, there is no tradition in Denmark for systematical communication about wishes for end-of-life care. The aim of the study is to adapt the ACP to a new contest and target group and determine the feasibility and acceptable recruitment rate and completeness of potential outcome measures for a future RCT.

A study of a complex intervention will be conducted to address all elements of an adapted ACP intervention in HF patients (NYHA class III, IV) and their relatives. Patients will be identified and recruited by HF specialist nurses or a cardiologist from the Department of Cardiology at North Zealand Hospital. The HF specialist nurses or the cardiologist will inform the patients about the study and obtain consent for the research staff to contact the patients by telephone. The patients will be further informed by the research staff and asked to fill out the baseline questionnaires. The patients will be asked to select the closest relatives who also will be offered participation. Included patients will receive an invitation with the date and time of their ACP meeting in their electronic patient record. They will be offered an ACP discussion which covers components e.g. symptom control, discussions on prognosis and illness limitations, and wishes for future and end-of-life care. Baseline and follow-up (4 and 12 weeks after the ACP meeting) will be made with disease-specific and generic questionnaires. Qualitative interview data will be obtained, and thematic analysis will uncover the patients, relatives and the clinician's perspectives and satisfaction with the intervention.

DETAILED DESCRIPTION:
Background Advance care planning (ACP) represents a way to fulfil patients' end-of-life preferences and wishes and the opportunity to improve the quality of life (QoL) for patients with life-limiting diagnoses and their relatives. ACP is advocated to improve end-of-life care for patients with heart failure (HF). The American Heart Association (AHA) has emphasized the importance of discussing with patients via ACP to better co-ordinate future healthcare based on the patient's values, preferences, and wishes, as well as their current clinical status such as their symptoms and QoL, prognosis and potential treatment options. It is important to discuss ACP not only when the HF is exacerbated, but also early in the disease process because a person's preferences may change over time. This is supported by the European Society of Cardiology (ESC) in their recently published guidelines for the diagnosis and treatment of acute and chronic HF. Here they state that proactive decisions and ACP with regard to palliative and end-of-life care should be regularly reviewed and documented. A recent systematic review and meta-analysis showed that ACP discussions improved QoL, patient satisfaction with end-of-life care and the quality of end-of-life communication for patients suffering from HF and could be most effective when the right timing, follow-up and involvement of important others was considered. Previous reviews had investigated the effectiveness of interventions to implement ACP. However, they did not investigate the impact of ACP on HF.

A Danish position statement on palliative care (PC) and advanced heart disease was recently published. The intention was to inform and influence policy and practice and focused on HF, increases the awareness of the need for PC care among patients with non-malignant diseases and inspires the process of implementing and organizing PC in advanced heart disease in Denmark and Internationally. In line with AHA this Danish position statement includes the importance of communication and ensuring ACP support. However, despite the growing emphasis on communication with HF patients and their relatives in Denmark, there is no tradition for systematical communication about wishes for end-of-life care in the Hf patients and their relatives.

This study has been designed through a systematic intervention development based on best current knowledge and our hypothesis is that ACP could be adapted and feasible in a danish healthcare population of HF patients, New York Heart Association (NYHA) Functional Classification III and IV. However, there are some uncertainties that need to be tested before we progress to a fully powered randomized controlled trial (RCT). Therefore, the aim of the study is to adapt the ACP intervention to a new contest and target group and determine the feasibility and acceptable recruitment rate and completeness of potential outcome measures for a future RCT.

Study design Implementing evidence-informed population health interventions in new contexts often requires adaptations. Therefore, an adaptation study of a complex intervention will be conducted to address all elements of the planned intervention to ensure that the intervention is feasible in HF patients and their relatives in the current context. The study will be conducted in a manner that increase external validity.

The methods regarding ACP discussions are adapted from a previous danish study. The inclusion criteria are based on the ESC guidelines according to patients with HF in whom PC and end-of-life care should be considered. To ensure a viable design, the existing model will be adapted and modified to our current context. The study will include 20 patients and their relatives with the purpose to test the feasibility and evaluate the intervention in our setting. Four new patients will be invited every month and the inclusion period is approximately expected to last 5 months. Criteria's will be agreed to provide a transparent decision process on readiness to progress to a fully powered RCT. Likewise, to identify where and to what extent the study design and/or intervention may need to be amended. There are three areas that need special attention; 1) how many HF patients will meet the inclusion criteria; 2) will the HF patients and their relatives accept and be engaged in the intervention; and 3) are the HF patients and their relatives able to complete the online survey. The study will be reported according to the CONSORT extension for pilot and feasibility trials.

Participants Patients ≥18 years with HF NYHA class III-IV in acute exacerbation who are admitted to the Department of Cardiology, North Zealand Hospital and fulfil the inclusion criteria will be asked to participate. The patients will be asked to select the closest relatives, who also will be offered participation.

Intervention The patient will be offered a intervention by the Department of Cardiology. The intervention covers a ACP discussion including symptom control. The intervention consists of a dialogue between the patient, the closest relative, a cardiologist, a PC physician and a HF nurse. Based on the ACP approach the North Zealand hospital have built a smartphrase for documentation in the electronic patients' records. The smartphase includes eight questions; 1. Introduction to the purpose of the ACP discussion; 2. Clarification of the closest relative(s); 3. Clarification of what the patient and the relatives know about the disease and its trajectory; 4. Clarification of what the most important things are to the patient to be able to do; 5. Clarification of the patient's and relatives' experiences of incurable disease and their preferences regarding end-of-life care; 6. Clarification of the patients' wishes and possibilities to level of treatment; 7. Clarification of the patient's wishes in preferred place of care and death; 8. Clarification of whether there is something the health professionals need to know in order to fulfill the patient's wishes at the preferred place of care and death. The intervention will be implemented on the basis of Detering et al. five factors for improving patient satisfaction with end-of-life care discussions: (1) using trained facilitators,(2) conducting a patient-centred discussion,(3) the involvement of the family,(4) correctly filing and communicating the ACP documentation with all parties, and (5) education of doctors in communicating ACP. A future plan will be made in collaboration by the patient, the relative, the cardiologist, the PC physician, and the HF nurse at the end of the ACP discussion. After the end of discussion, the patient's wishes and future preferences will be documented in their individual patient record. With the patient's acceptance their GP will receive a copy of the ACP document.

Evaluation To identify potential primary outcomes for a future effect study and provide limited efficacy testing, data will be collected in a structured way to investigate changes in the patient-reported outcome measurements (PROMs), including assessments of symptoms, health-related quality of life (HRQoL) and caregiver burden.

All questionnaires will be sent electronically to the patients and the relatives through REDCap. This is a secure web application for building and managing online surveys and databases. The research staff will support all patients and relatives not used to filling out questionnaires in electronically systems.

Patient, relatives and clinician satisfaction Qualitative interview is a well-suited method when knowledge is wanted on how informants describe their experiences. After the ACP meeting an evaluative semi-structured telephone interview will be conducted with all participants to obtain a deeper understanding of their experiences. The interviews will take place maximum two weeks after the ACP meeting. All interviews will be performed by research staff. The interviews will be guided by questions based on an interview guide. Each interview will be initiated with an open question on the patient's disease trajectory followed by their recollection of positive or negative experiences with the ACP meeting.

A qualitative focus group-interview will be conducted with the clinicians involved after study completion where the clinician's satisfaction with the intervention will be investigated. All interviews will be recorded, transcribed. All interviews with patients will be rendered anonymous.

Analyses Statistical analysis will be performed, considering the selection of appropriate analysis methods. For self-reported outcome scores, continuous data will be checked for normality and presented as mean ± standard deviation (SD). Frequencies will be expressed as percentages. Mean difference will be determined to investigate change in outcomes from baseline to follow-up time points. Due to the small numbers planned to be included in the present study only simple statistics will be applied. Effect size will be estimated with Cohen's d; values of 0.3, 0.5 and 0.8 will be interpreted as small, medium and large effect sizes respectively. All analyzes will be performed in SAS 9.4.

Thematic analysis will be used to analyze all the interviews and was chosen to extract data, and to identify and report patterns. NVivo will be used to code and retrieve data.

Strengths The ACP intervention has proved to be feasible and successful in different patient populations and has specific strengths. It includes both patients and their relatives and has been adapted to be HF specific and the intervention includes individually tailored provision of and discussion of prognostic information and end-of-life care preferences and wishes. This study, also, has methodological strengths. It is a study of a complex intervention where the process is dynamic, iterative, creative, open to change and forward looking to future evaluation and implementation if proven to be successful. Finally, the study will be the key to inform of the feasibility and design of a full-scale RCT.

Limitations The proportion of patients who participate in the trial will be documented. However, it is likely that there will be systematic differences between those who participate in the ACP trial and those who do not want to participate. Also, it is unavoidable that in conducting a study involving patients with incurable HF, a number of participants may die before follow-up data can be collected or wish to withdraw from the study before completion.

Disclosures and dissemination The study will be performed in accordance with the Declaration of Helsinki and will be registered on clinicaltrials.gov. It has been approved by the Danish Data Protection Agency (P-2020-790) and assessed by the Danish Ethics Committee (H-20041951).

Results from the study will be reported through oral presentations at national and International meetings and publication in international journals. The results will be published according to the 'CONSORT Statement' (www.consort-statement.org).

Funding The study is supported by Aase og Ejnar Danielsens foundation and the Department of Cardiology and the Department of Oncology and Palliative Care at the North Zealand Hospital.

ELIGIBILITY:
Inclusion criteria - patients:

* At least 18 years of age
* Able to speak and understand Danish
* Not expected to die within 1 month assessed by a cardiologist or a heart failure specialist nurse
* Cognitively able to participate in the intervention

Disease specific criteria - patients (minimum two must be fulfilled):

* Classified as being in NYHA III-IV by a cardiologist or heart failure specialist nurse and documented in the patient record.
* Progressive functional decline (physical and mental) and dependence in most activities of daily living based on clinical assessment by a cardiologist or a heart failure specialist nurse.
* Severe symptoms despite optimal pharmacological and non-pharmacological treatment assessed by a cardiologist or a heart failure specialist nurse.
* Two or more acute episodes that required admission to hospital over the last 6 months including the current admission.
* Heart transplantation and mechanical circulatory support (MCS) ruled out.
* Cardiac cachexia assessed clinically defined as a 'complex metabolic syndrome associated with underlying illness and characterized by loss of muscle with or without loss of fat mass'.
* Clinically judged by a cardiologist, palliative specialist or heart failure specialist nurse to have a life expectancy within 1-12 month.

Inclusion criteria - caregivers:

• At least 18 years of age

Exclusion criteria:

* Unable to speak or communicate in Danish
* Cognitively unable to participate to collaboration and complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life | Baseline, after 4 and 12 weeks
  • The European Organisation for Research and Treatment of Cancer Quality of life - Questionnaire - (EORTC QLQ-C15-PAL) to assess several physical and psychosocial aspects of the patient's health-related quality of life. Each question is rated on a Likert scale from 1 (not at all) to 4 (very much) excluding global health status, which is rated from 1 (very poor) to 7 (excellent).
Change in Quality of life and heart related symptoms | Baseline, 4 and 12 weeks
  • HeartQol to assess health-related quality of life in patients with heart disease. Each question is scored on a 4-point Likert scale from 0-3. The higher score, the less the respondent is bothered by his heart problem, which means a higher quality of life.
Change in Fatique | Baseline, 4 and 12 weeks
  • Multidimensional Fatigue Interventory (MFI-20) to determining the quality and patterns of sleep. The items are rated on agreement with statements (Yes, that is true - No, that is not true) covering five dimensions of fatigue. Range 4-20. Higher scores indicate greater fatigue.
Change in Anxiety and depression | Baseline, 4 and 12 weeks
  • Hospital Anxiety and Depression Scale (HADS) to assess anxiety and depression in medically ill patients. A 14 items in two sub-scales (anxiety: HADS-A; depression: HADS-D). Total subscale scores range: 0-21. Both subscale scores can be interpreted as follows: 0-7 points is considered within normal range, 8-10 is suggestive of the mood disorder, ≥8 indicating probable presence of the mood disorder.

SECONDARY OUTCOMES:
Use of healthcare system-patients' assessment | During the past 12 months from intervention.
  • Clinical information collected from patients' records regarding number of hospitalizations and days spent in hospital.
Change in Dyadic coping-patients and caregivers' assessment | Baseline, 4 and 12 weeks
  • Dyadic Coping inventory, will be used to assess how patients and relatives manage stress together concerning decision making and giving support to each other. A 37-item instrument designed to measure perceived communication and dyadic coping that occurs in close relationships when one or both partners are stressed. The items are rated on a 5-point Likert scale from ("very rarely") to 5 ("very often").
Change in Caregiver burden -caregivers' assessment | Baseline, 4 and 12 weeks
  • Zarit Burden Interview measures subjective caregiver burden. It examines burden associated with functional/behavioral impairments and the home care situation. A 22-item instrument rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater caregiver burden. A score of 17 or more is considered high burden.
Change in Health-related quality of life-patients and caregivers' assessment | Baseline, 4 and 12 weeks
  • RAND 36-Item Short Form Health Survey version 1.0 (SF-36), will be used to assess health-related quality of life. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Satisfaction with the intervention - interview with patients and caregivers | Maximum 2 weeks after the ACP intervention
  • The patients and caregivers will be invited for an semi-structured interview.
Satisfaction with the intervention - interview with healthcare professionals | Through study completion, an average of 7 month
  • Healthcare professionals involved in the study will be invited for an semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Lykke, Postdoc, Principal Investigator — Department of Oncology and palliative Care and the Department of Cardiology, North Zeeland Hospital; Camilla Lykke, Postdoc, Study Director — Department of Oncology and palliative Care and the Department of Cardiology, North Zeeland Hospital
Locations (1):
- Department of Cardiology, North Zeeland Hospital, Hillerød, Denmark

REFERENCES:
- [Derived] Roin T, Jurlander B, Juhl GI, Dieperink KB, Sjogren P, Bergenholtz H, Zwisler AD, Kurita GP, Larsen S, Tonder N, Hoyer LV, Lykke C. Taking a stand, ready or not: navigating sensitive end-of-life care conversations in patients with end-stage heart failure. Eur J Cardiovasc Nurs. 2025 Apr 11;24(3):401-410. doi: 10.1093/eurjcn/zvae170. PMID 39762160